CLINICAL TRIAL: NCT02873039
Title: Correlation Between Estimated Right Atrial Pressure and BNP in Pulmonary Hypertension (CRAB-PH)
Brief Title: Correlation Between Estimated Right Atrial Pressure and BNP in Pulmonary HTN (CRAB-PH)
Acronym: CRAB-PH
Status: Completed | Type: Observational
Sponsor: Louisiana State University Health Sciences Center in New Orleans (Other)
Responsible Party: Principal Investigator, Matthew Lammi, Assistant Professor of Medicine, Louisiana State University Health Sciences Center in New Orleans
Other Study IDs: IRB 9403
Record Dates: First submitted 2016-08-12; First posted 2016-08-19 (Estimated); Last update posted 2021-09-10 (Actual); Status verified 2021-09

CONDITIONS: Pulmonary Hypertension
MeSH Terms: conditions — Hypertension, Pulmonary

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

SUMMARY:
Over the past decade, advancements in therapies available for pulmonary hypertension (PH) have increased life expectancy for those who qualify and receive treatment. Yet, prognostication of these patients has remained a clinical dilemma. The application of the REVEAL registry predictive algorithm provides information about estimated 1-year survival but since invasive measurements from a right heart catheterization cannot easily be repeated, it is not feasible to continually use this longitudinally to assess the disease burden. Simple tests such as BNP has been shown to be very clinically relevant in short -term and long term prognostication and seems to correspond well to the right ventricular failure. Elevated right atrial pressures, and its estimation via IVC measurements predict poor survivorship in a recent retrospective analysis. As clinical measurement of jugular venous pressure is becoming less reliable, we aim to bring point- of-care ultrasound to the outpatient setting. Point of care ultrasound is widely used in the Emergency Department and Intensive Care Unit settings. By measuring estimated right atrial pressure (eRAP) via Inferior Vena Cava (IVC) measurements at outpatient clinic visits we aim to find a correlation with the existing and widely used B-type Natriuretic Peptide (BNP), that is collected at each visit as a part of regular care. These measurements can be followed longitudinally and may aid in prognostication. Data will be collected over the period of 1 year at clinic visits. A composite endpoint (including death, hospitalizations for PH, addition of new PH specific therapy after a stabilization period of 3 months, lung transplant or atrial septostomy) will separately be collected. At the end of the data collection period, clinical data only will be collected for a additional 2 years via phone correspondence, chart review or at regular PH clinic visits.

DETAILED DESCRIPTION:
Pulmonary hypertension patients who choose to participate:

Written informed consent will be obtained for the study. Patients must sign the informed consent before participating in any study related procedures.

* All inclusion and exclusion criteria will be reviewed.
* Demographic history will be recorded.
* Vital signs will be performed.
* A medication history will be taken.
* A smoking history will be recorded.
* BNP levels will be measured as a part of usual care at PH visits.
* Ultrasonographic measurements will be performed at the clinic visit.
* Ultrasonographic measurements:

IVC Measurements

* Performed in the subcostal view in supine position.
* Images will be captured in a video format.
* Maximal IVC diameter 1 to 2 cm from the junction of the right atrium and the IVC at end-expiration just proximal to the junction of the hepatic veins. The IVC collapsibility index to give an estimate of RAP.
* Inspiratory collapse of > 50% or < 50% will be ascertained based on the measurements.

Jugular Vein Measurements

* Patient will be placed in 45° position
* Longitudinal images will be obtained of the right jugular vein.
* Location of tapering of the jugular vein is measured, and distance from the sternal angle is recorded as ultrasound-measured jugular venous pressure (JVP).

Clinical Worsening Outcomes

• At each visit during year 1, and then every 6 months for years 2-3, clinical worsening events will be captured. These events are defined as:

* Death
* PH-related hospitalization
* Lung transplant
* Atrial septostomy
* Functional Class worsening and step up in therapy

Study Timing

* Enrollment of patients for a period of 1 year. Subsequently, no more patients will be enrolled. Patients who are enrolled will be followed clinically without further study-related testing at their regular clinic visits after completion of year 1.
* All patients enrolled will have ultrasonographic measurements of IVC and jugular veins at each clinic visit for 1 year.
* Data collection regarding meeting clinical worsening end points and BNP levels will be collected at the regular clinic visits at year 2 and 3 of the study.
* If patients are lost to follow up at clinics (including year-1), telephone correspondence, social security database review or chart review at 6-month intervals will be performed to determine vital status and see if they have met any clinical worsening endpoints.
* Study will close after the final patient has completed 3-years of follow up.

ELIGIBILITY:
Inclusion Criteria:

* Age > 18
* Clinical diagnosis of pulmonary hypertension
* BNP levels measured on day of clinic visit

Exclusion Criteria:

* Pregnant females
* Inability to lay flat for the ultra-sonographic measurements

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients who present to the University Medical Center with a clinical diagnosis of pulmonary hypertension.
Sampling Method: Non-Probability Sample
Enrollment: 90 (Actual)
Dates: Start 2016-07 (Actual); Primary Completion 2018-05 (Actual); Study Completion 2020-07 (Actual)

PRIMARY OUTCOMES:
Number of patients who show a relationship between inferior vena cava (IVC) measurements, eRAP and BNP using ultrasound. | 1 year
  To accomplish this objective, ultrasonographic measurements of the IVC and jugular veins will be performed at each visit, which can be easily measured longitudinally to establish a relationship with BNP.

SECONDARY OUTCOMES:
Time to Clinical worsening | 2 years
  Any outcome measure that indicates the patient is clinically worse than the previous visit will be considered in the assessment of time to clinical worsening. The 2 year follow-up period will assess:
  1. All-cause death
  2. Need for atrial septostomy
  3. Need for lung transplant
  4. Hospitalization for PH
  5. Worsening functional class (or no improvement from functional class 4) and need for additional PH therapies after a period of initial clinical stabilization of 3 months.
  These outcomes will all be used in the determination of disease progression.

CONTACTS AND LOCATIONS:
Overall Officials: Matthew R Lammi, MD, MSCR, Principal Investigator — Louisiana State University Health Sciences Center - New Orleans
Locations (1):
- University Medical Center - New Orleans, New Orleans, Louisiana, United States

IPD SHARING:
Plan to Share IPD: No
Individual Participant Data (IPD) will not be made available.

REFERENCES:
- [Derived] Samant S, Tran HV, Uddo RB, deBoisblanc BP, Saketkoo LA, Saito S, Helmcke FR, Lammi MR. Use of Handheld Ultrasound to Estimate Right Atrial Pressure in a Pulmonary Hypertension Clinic. Ann Am Thorac Soc. 2022 Feb;19(2):179-185. doi: 10.1513/AnnalsATS.202101-092OC. PMID 34214012